CLINICAL TRIAL: NCT06832969
Title: A Clinical Study on Verifying the Cryoablation Technique for Peripheral Lung Malignancies Under Bronchoscopy Guidance
Brief Title: A Clinical Study of the Cryoablation Technique for Peripheral Lung Malignancies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Li Shiyue, Professor, Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cryobiopsy-lung-cancer
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer Patients
MeSH Terms: interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cryoablation (Experimental): Lung cancer patients undergo treatment for peripheral malignant lung tumors using cryoablation technology under the guidance of bronchoscopy.
  Interventions: Procedure: cryoablation

INTERVENTIONS:
Procedure: cryoablation — Lung cancer patients undergo treatment for peripheral malignant lung tumors using cryoablation technology under the guidance of bronchoscopy.

SUMMARY:
To assess the safety and effectiveness of bronchoscopy-guided cryoablation with cold verification for peripheral lung malignancies.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥ 18 years, with no gender restrictions; (2) Diagnosed as having peripheral lung cancer, with the maximum diameter of the tumor being ≤ 3 cm and the number of tumors being ≤ 3; (3) The lesion intended for ablation is evaluated as feasible for bronchoscopy-guided cryoablation therapy; (4) The subject refuses or is deemed unsuitable for radiotherapy/chemotherapy, or has no response to previous radiotherapy/chemotherapy, or has disease progression after radiotherapy/chemotherapy; (5) Assessed as ineligible for surgery or refuses surgery and radiotherapy, consents to receive initial ablation treatment and signs the informed consent form.

Exclusion Criteria:

* (1) Diffuse lesions in both lungs where ablation therapy fails to improve the condition; (2) Examinations within one month prior to the operation reveal the presence of hilar lymph node metastasis or extrapulmonary metastasis (except for cases where extrapulmonary metastasis has been controlled through local treatment); (3) Existence of contraindications for bronchoscopy, or inability of the patient to tolerate or cooperate with bronchoscopy; (4) Severe bleeding tendencies or uncorrectable coagulation dysfunctions (prothrombin time > 18 seconds, prothrombin activity < 40%); (5) Platelet count < 70×109/L, or discontinuation of anticoagulant and/or antiplatelet drugs less than one week before ablation (except for the prophylactic use of low-molecular-weight heparin before the operation); (6) Severe impairment of lung function with a maximum ventilation volume < 40%; (7) Concurrent presence of other tumors with extensive metastasis and an expected survival period of less than 3 months; (8) Poor overall condition (multiple metastases throughout the body, severe infection, high fever), infectious and radiation-induced inflammation around the lesion, obvious cachexia, severe dysfunction of important organs, severe anemia and short-term uncorrectable nutritional and metabolic disorders; (9) Eastern Cooperative Oncology Group (ECOG) performance status score > 2; (10) The lesion to be ablated has received radiotherapy within the past 6 months; (11) Active hepatitis B, active hepatitis C, human immunodeficiency virus (HIV) infection history (known positive for HIV1/2 antibodies), or other active infections that are judged by the researcher to potentially affect the patient's treatment; (12) Accompanied by epilepsy, history of mental illness or cognitive impairment; (13) Pregnant or lactating women, as well as male or female patients who plan to have children or become pregnant during the trial; (14) Participation in any other clinical trials within 3 months before signing the informed consent (excluding non-interventional studies); (15) Other circumstances deemed by the researcher as inappropriate for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete Ablation Rate | 6 months after biopsy
  It refers to the proportion of subjects in whom the major lesion remained completely ablated six months after the entire ablation procedure, as a percentage of all evaluable subjects who underwent cryoablation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakaji H, Niimi A, Matsuoka H, Iwata T, Cui S, Matsumoto H, Ito I, Oguma T, Otsuka K, Takeda T, Inoue H, Tajiri T, Nagasaki T, Kanemitsu Y, Chin K, Mishima M. Airway remodeling associated with cough hypersensitivity as a consequence of persistent cough: An experimental study. Respir Investig. 2016 Nov;54(6):419-427. doi: 10.1016/j.resinv.2016.06.005. Epub 2016 Jul 31. PMID 27886853